CLINICAL TRIAL: NCT05801458
Title: Evaluation of Resin Composite Posterior Restorations Using Modeling Resin Insertion Technique Versus Conventional Composite Placement Technique in Class I Lesions: Randomized Clinical Trial
Brief Title: Evaluation of Resin Composite Posterior Restorations Using Modeling Resin Insertion Technique in Class I Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ahmed Mahmoud Mohamed, Operator, main investigator and corresponding author, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Modeling Resin
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Class I Composite Restorations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modeling Resin Insertion Technique (Experimental): Resin Composite (Tetric® N-Ceram Nano-hybrid incremental composite) / Wetting Agent (Modeling Resin, Bisco)
  Interventions: Procedure: Modeling Resin Insertion Technique
- Conventional Resin Composite Incremental Placement Technique (Placebo Comparator): Conventional resin composite incremental placement technique (Tetric® N-Ceram Nano-hybrid incremental composite)
  Interventions: Procedure: Conventional resin composite Incremental Placement Technique

INTERVENTIONS:
Procedure: Modeling Resin Insertion Technique — One drop of modeling resin will be dispensed into a clean mixing well. Following the placement of the resin composite into the prepared site, a composite instrument (round-ended plugger with a diameter of 2 mm) will be dipped into the modeling resin. With modeling resin on the instrument, the resin composite is sculpted and manipulated to the desired shape. This will be repeated with each increment. Each increment will be polymerized for 20 sec with a LED light-curing unit.
  Arms: Modeling Resin Insertion Technique
Procedure: Conventional resin composite Incremental Placement Technique — A three-step etch-and-rinse adhesive system will be used according to the manufacturer's instructions. 37.5% phosphoric acid (Kerr Co, Orange, CA, USA) will be applied to the enamel and dentin for a period of 30 s and 15 s, respectively. Subsequently the cavities will then be rinsed with an air/water spray for 15 s. A layer of primer will be applied to the dentin for 30 sec, afterward gentle air-drying for 5 sec. Then, the bond (AdheSE adhesive) will be applied on the enamel and dentin and light cured with a LED curing unit for about 30 sec. Tetric N-Ceram will then be applied using an incremental filling technique, each increment will not exceed 2mm in thickness. Each increment will be polymerized for 20 sec with a LED light-curing unit.
  Arms: Conventional Resin Composite Incremental Placement Technique

SUMMARY:
Evaluation of Resin Composite Posterior Restorations Using Modeling Resin Insertion Technique versus Conventional Composite Placement Technique in Class I Lesions: Randomized Clinical Trial

DETAILED DESCRIPTION:
Statement of the problem In a restorative procedure, an important objective is to obtain restorations with smooth surfaces. Surface roughness has a major influence on plaque accumulation, secondary caries, and gingival irritation. Further, it may directly influence wear behavior and the marginal integrity of composite restorations. A roughened surface of a resin composite restoration is also likely to be stained by exogenous sources, such as coffee, tea, or red wine, leading to the discoloration of the material.

One of the main drawbacks of sculpting composite restorations is that some materials are sticky, reducing the ease of handling and insertion of the material into the tooth cavity. Some materials readily adhere to the composite instruments; thus, limiting reestablishment of the shape and anatomical contour of the tooth. As a result, the application of lubricants on the composite instrument such as modeling liquids/resins between the layers of composite have been proposed.

Rationale Modeling resins can be directly applied between the layers using a brush or can be used as a lubricant on manual instruments. In both the aforementioned techniques, the ease of instrumentation during the placement of esthetic restorations is superior, compared to the traditional restorative techniques. Moreover, any pores or gaps on the surface of the composite placed by means of the layering technique can be easily resolved. Hence, the modeling resin facilitates the reduction of defects in the body of the restoration and aids in improving the mechanical properties.

Although these methods are widely used, a potential shortcoming is that these techniques may adversely affect the physical and surface properties of the resin composite. However, it is unknown whether different compositions of adhesives or modeling agents may affect the surface microhardness, surface roughness, and color stability of composites over time.

ELIGIBILITY:
Inclusion Criteria:

Participants:

1. Adult Patients (25-45).
2. Good oral hygiene (plaque index score 0 or 1).
3. Absence of damaging habits (e.g. bruxism, nail biting, tooth clenching and mouth breathing).

Teeth:

1. Vital teeth with a normal appearance and morphology.
2. Primary carious lesions in molar teeth.

Exclusion Criteria:

Participants:

1. Patients with bad oral hygiene.
2. Patients with known allergic or adverse reaction to the tested materials.
3. Any uncontrolled systemic disease, pregnant or lactating women and any patient incapable to be present at recall follow up visits.

Teeth:

1. Non-vital, fractured, or cracked teeth.
2. Teeth with secondary caries or in need of replacement of existing restorations.
3. Defective restorations adjacent to or opposite the tooth restored in the study.
4. Rampant caries, atypical extrinsic staining of teeth.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Marginal Discoloration at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to delta (Immediate replacement necessary).

SECONDARY OUTCOMES:
Change from baseline in Marginal Integrity at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to delta (Immediate replacement necessary).
Change from baseline in Color Match at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to charlie (outside the acceptable range).
Change from baseline in Surface Roughness at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to delta (Immediate replacement necessary).
Change from baseline in Anatomic form (wear) at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to delta (Immediate replacement necessary).
Change from baseline in Retention of Restoration at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to charlie (complete loss of restoration).
Change from baseline in Secondary Caries at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to bravo (Caries contiguous with the restoration margin).
Change from baseline in Postoperative Sensitivity at 3,6,12 & 18 months | T1: 3 months • T2: 6 months • T3: 12 months • T4: 18 months
  Modified US Public Health Service criteria. Possible scores range from alpha (Excellent) to delta (Immediate replacement necessary).

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Abdelhamid, Professor-Cairo University, Study Director — Cairo University

REFERENCES:
- [Background] Barcellos DC, Pucci CR, Torres CR, Goto EH, Inocencio AC. Effects of resinous monomers used in restorative dental modeling on the cohesive strength of composite resin. J Adhes Dent. 2008 Oct;10(5):351-4. PMID 19058680
- [Background] Bayraktar ET, Atali PY, Korkut B, Kesimli EG, Tarcin B, Turkmen C. Effect of Modeling Resins on Microhardness of Resin Composites. Eur J Dent. 2021 Jul;15(3):481-487. doi: 10.1055/s-0041-1725577. Epub 2021 May 26. PMID 34041724
- [Background] Burke FJ, Crisp RJ, James A, Mackenzie L, Pal A, Sands P, Thompson O, Palin WM. Two year clinical evaluation of a low-shrink resin composite material in UK general dental practices. Dent Mater. 2011 Jul;27(7):622-30. doi: 10.1016/j.dental.2011.02.012. Epub 2011 Apr 22. PMID 21514654
- [Background] Dionysopoulos D, Papadopoulos C, Koliniotou-Koumpia E. The evaluation of various restoration techniques on internal adaptation of composites in class v cavities. Int J Biomater. 2014;2014:148057. doi: 10.1155/2014/148057. Epub 2014 Oct 2. PMID 25349611
- [Background] Furuse AY, Gordon K, Rodrigues FP, Silikas N, Watts DC. Colour-stability and gloss-retention of silorane and dimethacrylate composites with accelerated aging. J Dent. 2008 Nov;36(11):945-52. doi: 10.1016/j.jdent.2008.08.001. Epub 2008 Sep 7. PMID 18778884
- [Background] He Z, Shimada Y, Tagami J. The effects of cavity size and incremental technique on micro-tensile bond strength of resin composite in Class I cavities. Dent Mater. 2007 May;23(5):533-8. doi: 10.1016/j.dental.2006.03.012. Epub 2006 May 24. PMID 16725190
- [Background] Ilie N, Kessler A, Durner J. Influence of various irradiation processes on the mechanical properties and polymerisation kinetics of bulk-fill resin based composites. J Dent. 2013 Aug;41(8):695-702. doi: 10.1016/j.jdent.2013.05.008. Epub 2013 May 21. PMID 23707645
- [Background] Jefferies SR. Abrasive finishing and polishing in restorative dentistry: a state-of-the-art review. Dent Clin North Am. 2007 Apr;51(2):379-97, ix. doi: 10.1016/j.cden.2006.12.002. PMID 17532918
- [Background] Kohler B, Rasmusson CG, Odman P. A five-year clinical evaluation of Class II composite resin restorations. J Dent. 2000 Feb;28(2):111-6. doi: 10.1016/s0300-5712(99)00059-7. PMID 10666968
- [Background] Munchow EA, Sedrez-Porto JA, Piva E, Pereira-Cenci T, Cenci MS. Use of dental adhesives as modeler liquid of resin composites. Dent Mater. 2016 Apr;32(4):570-7. doi: 10.1016/j.dental.2016.01.002. Epub 2016 Feb 3. PMID 26850844
- [Background] Nahsan FP, Mondelli RF, Franco EB, Naufel FS, Ueda JK, Schmitt VL, Baseggio W. Clinical strategies for esthetic excellence in anterior tooth restorations: understanding color and composite resin selection. J Appl Oral Sci. 2012 Mar-Apr;20(2):151-6. doi: 10.1590/s1678-77572012000200005. PMID 22666829
- [Background] Rees JS, Jagger DC, Williams DR, Brown G, Duguid W. A reappraisal of the incremental packing technique for light cured composite resins. J Oral Rehabil. 2004 Jan;31(1):81-4. doi: 10.1046/j.0305-182x.2003.01073.x. PMID 15125602
- [Background] Rosa WL, Piva E, Silva AF. Bond strength of universal adhesives: A systematic review and meta-analysis. J Dent. 2015 Jul;43(7):765-76. doi: 10.1016/j.jdent.2015.04.003. Epub 2015 Apr 14. PMID 25882585
- [Background] Sedrez-Porto JA, Munchow EA, Cenci MS, Pereira-Cenci T. Translucency and color stability of resin composite and dental adhesives as modeling liquids - A one-year evaluation. Braz Oral Res. 2017 Jul 3;31:e54. doi: 10.1590/1807-3107BOR-2017.vol31.0054. PMID 28678973
- [Background] Sirin Karaarslan E, Bulbul M, Yildiz E, Secilmis A, Sari F, Usumez A. Effects of different polishing methods on color stability of resin composites after accelerated aging. Dent Mater J. 2013;32(1):58-67. doi: 10.4012/dmj.2012-045. PMID 23370871
- [Background] Suneelkumar C, Harshala P, Madhusudhana K, Lavanya A, Subha A, Swapna S. Clinical performance of class I cavities restored with bulk fill composite at a 1-year follow-up using the FDI criteria: a randomized clinical trial. Restor Dent Endod. 2021 Apr 16;46(2):e24. doi: 10.5395/rde.2021.46.e24. eCollection 2021 May. PMID 34123760
- [Background] Tanaka A, Nakajima M, Seki N, Foxton RM, Tagami J. The effect of tooth age on colour adjustment potential of resin composite restorations. J Dent. 2015 Feb;43(2):253-60. doi: 10.1016/j.jdent.2014.09.007. Epub 2014 Sep 19. PMID 25242100
- [Background] Tuncer S, Demirci M, Tiryaki M, Unlu N, Uysal O. The effect of a modeling resin and thermocycling on the surface hardness, roughness, and color of different resin composites. J Esthet Restor Dent. 2013 Dec;25(6):404-19. doi: 10.1111/jerd.12063. Epub 2013 Oct 31. PMID 24172016
- [Background] van Dijken JW, Pallesen U. A 7-year randomized prospective study of a one-step self-etching adhesive in non-carious cervical lesions. The effect of curing modes and restorative material. J Dent. 2012 Dec;40(12):1060-7. doi: 10.1016/j.jdent.2012.08.017. Epub 2012 Sep 3. PMID 22955004